CLINICAL TRIAL: NCT04788979
Title: The Adjunctive Use of Systemic Melatonin Therapy in the Treatment of Periodontitis Associated With Obesity (Clinical and Immunological Study).
Brief Title: The Adjunctive Use of Melatonin Therapy in the Treatment of Obese Periodontitis Patients (Clinical and Immunological Study).
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, sami Hussam, Doctor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: melatonin and periodontitis
Record Dates: First submitted 2021-02-28; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Melatonin; Tablets

STUDY DESIGN:
Intervention Model Description: The subjects included in the study were the following:
  1-control group:20 subjects (healthy) 2-30 obese periodontitis patients.dont take melatonin 3-30 obese periodontitis patients taking melatonin
Who Masked: Investigator
Masking Description: self investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Melatonin 5Mg Oral Tablet — 1. control without treatment
  2. obese periodontitis patients treated only by scaling and root planning
  3. obese periodontitis patients treated with scaling and root planning with daily dietary supplementation of 5 mg melatonin (NOW-USA)

SUMMARY:
To evaluate the effect of adjunctive systemic administration of melatonin to mechanical non- surgical periodontal therapy in obese patients with periodontitis.

DETAILED DESCRIPTION:
Periodontitis defined as destruction of periodontal tissue caused by specific microorganisms resulting of pocket formation, recession and mobility.Obesity known to increase the host tolerance by influencing the immune and inflammatory mechanisms in a way that inflammatory tissue destruction is predisposed and leave a person at high risk of developing periodontitis.the relationship between periodontitis and obesity has been reported in several epidemiological and experimental studies.

Obesity can be a higher trigger of chronic stress , stress and how a person copes with stress has been shown to increase the risk of periodontitis.several studied have shown that preserving of normal weight by maintaining regular physical exercise is linked with a lower incidence of periodontitis.

As a matter of truth , overweight and obese individuals are more than twice as likely to have periodontitis compared to normal healthy persons. It has been suggested that obesity decreased the blood flow to periodontal tissue, enabling the development of periodontal disorders. The blood vessels of obese subjects demonstrate a thickening in the inner wall of arteries that reduce the flow of blood into periodontium. The adipocytes produce various active molecules called adipokines involving (TNF- α, IL-6, leptin, adiponectin and others). These compound secrete various molecules of reactive oxygen species (ROS) that lowered antioxidant enzymes activity like (superoxide dismutase, catalase, glutathione and others). Thus modulating the effect of adipokines can lower the pathogenicity of periodontitis by reducing the effect of oxidative stress.

Oxidative stress appear to be the main link between obesity and periodontitis and can aggravates pro-inflammatory pathways frequent in both pathologies. Regarding the significance of oxidative stress in pathologies of both periodontitis and obesity, several antioxidants play an amazing role as a preventive and therapeutic measures for both diseases. Multiple studies had a greater evidence toward melatonin which have an active antioxidant properties , which is an indolamine produced mainly by pinealocytes. It has been documented that salivary melatonin were significantly decreased in patients with periodontal disease, indicated that melatonin may act as a biomarker for periodontal diagnosis and can be used as a possible therapeutic agent in various periodontal diseases.

It is indicated that adjunctive use of melatonin in combination with non-surgical scaling and root planning for 3 weeks can lead to improvement of clinical periodontal parameters in diabetic patients. It was demonstrated that daily dietary supplementation with 3mg melatonin tablet for 4 weeks along with scaling and root planning significantly reduced the oxidative stress in periodontitis patients.

similarly , significant reduction in gingival inflammation when melatonin administrated locally as adjunctive measure to standard periodontal therapy. Melatonin promote bone formation by activating type 1 collagen fibers in osteoblast and enhancing the genetic expression of bone sialoprotein , alkhaline phosphates, osteopontien and osteocalcine and downregulate the RANKL mediated osteoclast formation and activation.

It had been reported that circulatory serum level of melatonin significantly reduced in obesity .Supplementation of antioxidants in conjunction with other treatment modalities such as dietary changes, behavioral changes, and drug therapy might be beneficial in treatment of obesity and associated inflammatory states ., as melatonin participated in homeostasis and metabolism of energy through activation of brown adipose tissue and enhance energy expenditure. furthermore, significant reduction in body weight along with adipose tissue deposit when melatonin were administrated in obese subjects was reported in. Multiple studies reported that melatonin significantly increase HDL level and decrease TG and HDL level in addition to increased cholesterol catabolism.

ELIGIBILITY:
Inclusion Criteria:The study involve three groups: the first one is control (healthy normal weight group).

The second one is experimental group which must have the following criteria:

1-latest sleep, obese patients diagnosed to have periodontitis with probing pocket depth ≥ 5mm, 2-patients able to follow the required instruction.

-

Exclusion Criteria:1-individuals having night work shifts. 2-patients wearing removable partial dentures and undergoing orthodontic treatment.

3-patient taking anti-inflammatory drugs, antibiotics, immunosuppressant or oral contraceptives since last 3 months.

4-paients with diabetic mellitus, liver diseases, autoimmune diseases and osteoporosis.

5-pregnant or lactating women. 6-cancer patient. 7-smoker patient.

-

Ages: 27 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
measurement of clinical periodontal parameters | 4 weeks
  1. plaque index
  2. gingival index
  3. bleeding on probing
  4. pocket depth
  5. relative attachment level all parameters are recorded by using periodontal probe.
measurement of biochemical markers in serum | 4 weeks
  1. measurement of receptor activator of nuclear KB receptor
  2. measurement of total antioxidant capacity
  3. measurement of melatonin level all markers are recorded by using Eliza

SECONDARY OUTCOMES:
measurement of lipid profiles in serum | 4 weeks
  cholesterol, triglycerides,HDL,LDL
measurement of BMI | base line visit
  multiple measurements will be aggregated to arrive at one reported value (e.g., weight and height will be combined to report BMI in kg/m^2).

CONTACTS AND LOCATIONS:
Locations (1):
- university of Baghdad, Baghdad, Iraq

REFERENCES:
- [Background] Gitto E, Aversa S, Reiter RJ, Barberi I, Pellegrino S. Update on the use of melatonin in pediatrics. J Pineal Res. 2011 Jan;50(1):21-8. doi: 10.1111/j.1600-079X.2010.00814.x. Epub 2010 Oct 1. PMID 21029156
- [Background] Andersen LP, Rosenberg J, Gogenur I. Perioperative melatonin: not ready for prime time. Br J Anaesth. 2014 Jan;112(1):7-8. doi: 10.1093/bja/aet332. No abstract available. PMID 24318695